CLINICAL TRIAL: NCT01843452
Title: Phase II Study of Concomitant Intensity-modulated Radiotherapy Combined to Capecitabine, Mitomycin and Panitumumab in Patients With Stage II-IIIB Squamous-cell Carcinoma of the Anal Canal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Oscar Matzinger, Senior Physician & senior lecturer, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV 20080214
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Carcinoma of Anal Canal
MeSH Terms: conditions — Anal Canal Carcinoma | interventions — Radiotherapy; Panitumumab; Mitomycin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine, mitomycin, panitumumab and radiotherapy (Experimental): RADIOTHERAPY: daily fraction dose of 1.8Gy , 5 days a week between day 1 and 45 Intensity modulated radiotherapy (IMRT), using a linac based facility or helical tomotherapy, is obligatory.
  The first treatment sequence consists of a total dose of 36 Gy in 20 daily fractions of 1.8 Gy on five days a week.
  The second treatment sequence consists of a total dose of 23.4 Gy in 13 daily fractions of 1.8 Gy on five days a week.
  PANITUMUMAB: 6 mg/kg IV over 60 min infusion on days 1, 15 and 29
  MITOMYCIN: 10 mg/m2 IV over 15 min infusion on days 1 and 29
  CAPECITABINE: 825 mg/m2 oral twice daily on days 1 to 45
  Interventions: Radiation: RADIOTHERAPY; Biological: PANITUMUMAB; Drug: MITOMYCIN; Drug: CAPECITABINE

INTERVENTIONS:
Radiation: RADIOTHERAPY — External beam radiotherapy (daily fraction dose 1.8Gy) on Monday through Friday starting on study day 1.
  * Days 1-28, dose of 36 Gy in 1.8 Gy/fraction (20 fractions) to the clinical target volume 1 (CTV1) including the primary tumor and involved lymph nodes and areas at risk for metastatic spread (which includes gross tumour volumes (GTV) and a 1-cm expansion, mesorectal space, inguinal, femoral, external iliac, internal iliac, and common iliac vessels).
  * Days 29-45, a boost dose of 23.4 Gy in 1.8 Gy/fraction (13 fractions) to the GTV.
Biological: PANITUMUMAB — 6 mg/kg IV administered over 60 min infusion on days 1,15 and 29.
Drug: MITOMYCIN — 10 mg/m2 IV administered over 15 min infusion on days 1 and 29.
Drug: CAPECITABINE — 825mg/m2 orally twice daily on study days 1 through 45.

SUMMARY:
There is increasing evidence of a role of EGFR, treatment with EGFR-inhibitors in anal cancer and synergies of EGFR-inhibitors with radiotherapy. Addition of the human anti-EGFR antibody Panitumumab to chemoradiotherapy seems therefore solidly justified. This trial investigates concurrent panitumumab/capecitabine/mitomycin concurrent to IMRT-radiotherapy. Treatment components used in this study have been selected on scientific rationale. The trial regimen should be feasible with acceptable toxicity and outcome similar to historic series.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

-To assess efficacy of treatment regimen composed of capecitabine, mitomycin, panitumumab, and radiotherapy in terms of locoregional control rate in patients with stage II-IIIB squamous-cell carcinoma of the anal canal.

Secondary:

* To further assess efficacy of this regimen based on complete response (CR) rate, colostomy-free survival, functional colostomy-free survival, overall survival (OS), and progression-free survival (PFS).
* To assess the tolerability and safety profile of this regimen.
* To assess the role of PET for staging and outcome prediction (for those patients who had PET following local standards).

ELIGIBILITY:
Inclusion Criteria:

* Histologically/pathologically confirmed squamous-cell carcinoma of the anal canal
* Stage II-IIIB (T2-4, N any, M0) disease
* Previously untreated disease
* Age ≥ 18 years at time of consent
* Life expectancy of at least 2 years
* ECOG performance status (PS) of 0 to 1
* Adequate bone marrow, liver and renal functions as assessed by the following laboratory requirements to be conducted within 14 days prior to registration.

  * Hemoglobin ≥ 90 g/l without transfusion requirement in the prior 4 weeks
  * Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  * ALT and AST ≤ 2.5 x ULN
  * Alkaline phosphatase < 4 x ULN
  * PT/PTT < 1.5 x ULN (patients who receive anticoagulation treatment with an agent such as warfarin or heparin will be allowed to participate; for patients on warfarin, close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at predose, as defined by the local standard of care.
  * Serum creatinine clearance ≤ 1.5 x ULN (≥ 60 ml/min calculated using the Cockcroft-Gault formula)
* Patients with stable HIV infection (i.e. undetectable viral load over the past 6 months while on HIV treatment and with CD4 count > 200 /ml) can be included.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Prior treatment with capecitabine or mitomycin
* Prior or concurrent chemotherapy, or any antitumoral hormonal therapy
* Prior treatment with panitumumab or other EGFR inhibitors
* Prior biologic therapy or immunotherapy, e.g. anti-TNF treatment etc.
* Less than 24 hours since prior granulocyte colony-stimulating factors
* Any other concurrent anticancer therapy, including experimental medications
* Receipt of any investigational agent within 4 weeks of study registration
* Concurrent alternative medicine, vitamin supplements unless approved by the investigator
* Prior radiation therapy to the pelvis
* Prior surgery for anal canal cancer except biopsy
* Evidence of metastatic disease
* Prior or concurrent malignancy other than the study disease unless treated with curative intent and with no evidence of disease
* Any of the following within 6 months prior to study drug administration: severe/ unstable angina (symptoms at rest), new onset angina (began within the last 3 months) or myocardial infarction, congestive heart failure, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Known active Hepatitis B or C
* Active clinically serious infection > NCI-CTCAE v4.0 grade 3
* Known or suspected allergy to panitumumab or any agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Symptomatic pulmonary fibrosis
* History of collagen vascular disease
* Other severe, acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate contraception during the course of the trial and three months after the completion of trial
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2-year locoregional control in patients, which is defined as the absence of locoregional recurrence 2 years after treatment start.

SECONDARY OUTCOMES:
Complete response (CR) rate | 5 years
  Tumor assessment will be done by the investigator according to the RECIST 1.1. criteria.
Colostomy-free survival | 2 and 5 years
  2-year colostomy-free survival (patients without colostomy two-years after treatment start).
Functional colostomy-free survival | 2 and 5 years
  2-year functional colostomy-free survival (patients without colostomy and without stool incontinence or other sphincter symptoms interfering with activities of daily life two years after treatment start, which correspond to grade 3 toxicity according to common toxicity criteria National Cancer Institute-Common Toxicity Criteria for Adverse Event (NCI-CTCAE) version 4.0.
Overall survival (OS) | 2 and 5 years
  2-year overall survival (proportion of patients alive two years after treatment start) and median overall survival (median of the interval (days) between treatment start and death for any cause).
Progression-free survival (PFS) | 2 and 5 years
  2-year PFS (proportion of patients progression-free two years after treatment start) and median PFS according to the RECIST 1.1 criteria. PFS is defined as the interval (days) between registration and the date of progression (based on the actual tumor assessment date), or death for any cause, whichever comes first. The death of a patient without a reported progression will be considered as an event on the date of death. Patients who have neither progressed nor died will be censored on the date of last evaluable tumor assessment. Patients who had no post-baseline assessments and did not have an event will be censored at the time of registration.
Tolerability and safety profile of this regimen. | Early (6 weeks after treatment) and late (up to 2 and 5 years after treatment).
  Toxicities will be assessed according to the NCI-CTCAE (version 4.0).
Role of PET for staging and outcome prediction. | 5 years
  Predictive value of PET for PFS. Comparison of PET for determination of complete response with radiologic response and clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Matzinger, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (4):
- Switzerland (4):
  - Inselspital, Bern
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Hôpital du Valais (RSV), Sion